CLINICAL TRIAL: NCT02474316
Title: A Prospective, Randomized, Multicenter, Open-label Study Evaluating HBeAg Seroconversion in HBeAg Positive CHB Patients on Treatment With NA Switched to Combined Therapy With Peginterferon Alfa-2a and NA for 48 Weeks
Brief Title: Combined Therapy With Peginterferon Alfa-2a With NA in NA-treated HBeAg Positive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing XIe, Director of infectious disease, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2015-03-25; First posted 2015-06-17 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PegINF plus nucleos(i)de analgoue (Experimental): Peginterferon alfa-2a 180μg /wk plus nucleos(t)ide analgoue (NA) 1 piece qd for 48 weeks
  Interventions: Drug: Peginterferon alfa-2a; Drug: nucleos(t)ide analgoue
- nucleos(t)ide analgoue (Active Comparator): nucleos(t)ide analgoue (NA) 1 piece qd for 48 weeks
  Interventions: Drug: nucleos(t)ide analgoue

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a 180ug/wk s.c for 48 weeks
  Other Names: Pegasys
  Arms: PegINF plus nucleos(i)de analgoue
Drug: nucleos(t)ide analgoue — nucleos(t)ide analgoue (NA) 1 piece p.o for 48 weeks

SUMMARY:
This is a prospective, randomized, multicenter, open-label study. After more than 24 weeks NA treatment, HBeAg positive CHB patients who achieved HBV DNA<1000copies/ml but HBeAb negative, will be randomized (1:1) into 2 study arms as follows:

Arm A: Peginterferon alfa-2a 180μg /wk plus NA 1 piece qd for 48 weeks Arm B: Entecavir 0.5mg qd for 48 weeks

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter, open-label study. After more than 24 weeks NA treatment, HBeAg positive CHB patients who achieved HBV DNA<1000copies/ml but HBeAb negative, will be randomized (1:1) into 2 study arms as follows:

Arm A: Peginterferon alfa-2a 180μg /wk plus NA 1piece qd for 48 weeks Arm B:NA 1 piece qd for 48 weeks

The primary endpoint: HBeAg seroconversion at week 48

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with age ≥18 and ≤65 years;
2. There should be evidences that HBsAg and HBeAg have been positive for more than 6 months with HBsAb and HBeAb negative before treated with Entecavir;
3. Treated with NA for more than 24 weeks and achieve HBV DNA<1000copies/ml with HBeAb negative;
4. Women without ongoing pregnancy or breast feeding and willing to take an effective contraceptive measure during the treatment
5. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. Co-infection with active hepatitisA, hepatitisC, hepatitisD and/or human immunodeficiency virus (HIV)
2. AFP>50ng/ml and/or evidence of hepatocellular carcinoma
3. Evidence of decompensated liver disease (Child-Pugh scores >5). Child-Pugh >5 means that, if one of the following 6 conditions is met, the patient has to be excluded:

   1. Serum albumin <35 g/L;
   2. Prothrombine time prolonged≥ 4 seconds or PTA < 60%;
   3. Serum bilirubin > 34 µmol/L;
   4. History of encephalopathy;
   5. Ascites
4. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia)
5. Pregnant or breast-feeding Women
6. ANC<1.5x 10^9/L or PLT<90x 10^9/L
7. Consuming alcohol in excess of 20g/day for women and 30g/day for men within 6 months prior to enrollment
8. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis that treated with antidepressant medication or a major tranquilizer at therapeutic doses respectively at any time prior to 3 months or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
9. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.)
10. History of esophageal varices bleeding or other evidence of esophageal varices bleeding or other symptoms consistent with decompensated liver disease
11. History of chronic pulmonary disease associated with functional limitation
12. History of severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases)
13. Hemodialysis patients or patients with renal insufficiency
14. History of a severe seizure disorder or current anticonvulsant use
15. Major organ transplantation or other evidence of severe illness, malignancy, or any other conditions, which would make the patient, in the opinion of the investigator, unsuitable for the study
16. History of thyroid disease poorly controlled on prescribed medications
17. Evidence of severe retinopathy or clinically relevant ophthalmologic disorder
18. History of other severe disease or evidence of other severe disease or any other illness or conditions that the investigator believe that patients are not suitable to join in the study
19. Immunomodulatory treatment (including interferon) or LDT within 1 year prior to the first dose of treatment
20. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve HBeAg seroconversion | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the HBeAg seroconversion in HBeAg positive CHB patients on treatment with Entecavir and with HBV DNA <1000copies/ml which will be measured by the number of participants who achieve HBeAg seroconversion

SECONDARY OUTCOMES:
Number of participants who achieve HBeAg loss | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve HBeAg seroconversion which will be measured by number of participants who achieve HBeAg loss
Number of participants who achieve HBsAg loss | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve HBsAg loss which will be measured by number of participants who achieve HBsAg loss
Number of participants who achieve HBsAg seroconversion | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve HBsAg seroconversion which will be measured by number of participants who achieve HBsAg seroconversion
HBsAg decline from baseline | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve HBsAg decline from baseline
Percentage of participants who achieve HBsAg <1000IU/mL | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the percentage of participants who achieve HBsAg<1000IU/mL
Percentage of of participants who achieve HBsAg <100IU/mL | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the percentage of of participants who achieve HBsAg<100IU/mL
Number of participants who achieve combined response I (defined as HBeAg seroconversion and HBV DNA<100000copies/mL) | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the combined response I which will be measured by number of participants who achieve combined response I
Number of participants who achieve combined response II (defined as HBeAg seroconversion and HBV DNA<1000copies/mL) | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the combined response II which will be measured by number of participants who achieve combined response II
Number of participants who achieve dural response I (defined as HBeAg seroconversion and HBsAg<1000IU/mL) | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the dural response I which will be measured by number of participants who achieve dural response I
Number of participants who achieve dural response II (defined as HBeAg seroconversion and HBsAg<100IU/mL) | at week 48
  To investigate whether the combined therapy with Peginterferon alfa-2a with Entecavir can improve the dural response II which will be measured by number of participants who achieve dural response II
Number of Participants with AE | at week 48
  Number of participants with adverse events as a measure of safety and tolerability
Number of Participants with SAE | at week 48
  Number of participants with SAEs as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Qing Xie, Study Chair — Ruijin Hospital
Locations (3):
- China (3):
  - The Third People's Hospital of Guilin, Guilin
  - Ruijin Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai

REFERENCES:
- [Result] Lai CL, Ratziu V, Yuen MF, Poynard T. Viral hepatitis B. Lancet. 2003 Dec 20;362(9401):2089-94. doi: 10.1016/S0140-6736(03)15108-2. PMID 14697813
- [Result] Trepo C, Chan HL, Lok A. Hepatitis B virus infection. Lancet. 2014 Dec 6;384(9959):2053-63. doi: 10.1016/S0140-6736(14)60220-8. Epub 2014 Jun 18. PMID 24954675
- [Result] Tassopoulos NC, Volpes R, Pastore G, Heathcote J, Buti M, Goldin RD, Hawley S, Barber J, Condreay L, Gray DF. Efficacy of lamivudine in patients with hepatitis B e antigen-negative/hepatitis B virus DNA-positive (precore mutant) chronic hepatitis B. Lamivudine Precore Mutant Study Group. Hepatology. 1999 Mar;29(3):889-96. doi: 10.1002/hep.510290321. PMID 10051494
- [Result] Marcellin P, Chang TT, Lim SG, Tong MJ, Sievert W, Shiffman ML, Jeffers L, Goodman Z, Wulfsohn MS, Xiong S, Fry J, Brosgart CL; Adefovir Dipivoxil 437 Study Group. Adefovir dipivoxil for the treatment of hepatitis B e antigen-positive chronic hepatitis B. N Engl J Med. 2003 Feb 27;348(9):808-16. doi: 10.1056/NEJMoa020681. PMID 12606735
- [Result] Chang TT, Lai CL, Kew Yoon S, Lee SS, Coelho HS, Carrilho FJ, Poordad F, Halota W, Horsmans Y, Tsai N, Zhang H, Tenney DJ, Tamez R, Iloeje U. Entecavir treatment for up to 5 years in patients with hepatitis B e antigen-positive chronic hepatitis B. Hepatology. 2010 Feb;51(2):422-30. doi: 10.1002/hep.23327. PMID 20049753
- [Result] Brouwer WP, Xie Q, Sonneveld MJ, Zhang N, Zhang Q, Tabak F, Streinu-Cercel A, Wang JY, Idilman R, Reesink HW, Diculescu M, Simon K, Voiculescu M, Akdogan M, Mazur W, Reijnders JG, Verhey E, Hansen BE, Janssen HL; ARES Study Group. Adding pegylated interferon to entecavir for hepatitis B e antigen-positive chronic hepatitis B: A multicenter randomized trial (ARES study). Hepatology. 2015 May;61(5):1512-22. doi: 10.1002/hep.27586. Epub 2015 Feb 27. PMID 25348661